CLINICAL TRIAL: NCT03659643
Title: Mild Cognitive Impairment, Use of qEEG as a Prognostic Marker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jon Snaedal (Other)
Collaborators: Ullevaal University Hospital (Other); Karolinska University Hospital (Other); Rigshospitalet, Denmark (Other); Zealand University Hospital (Other); Haukeland University Hospital (Other); Kavli Research Foundation, Bergen Norway (Unknown)
Responsible Party: Sponsor-Investigator, Jon Snaedal, Professor in Geriatric Medicine, Landspitali University Hospital
Organization: Landspitali University Hospital (Other)
Other Study IDs: NORD-MCI
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI; Alzheimer´s disease; Lewy Body Dementia; EEG
MeSH Terms: conditions — Cognitive Dysfunction; Lewy Body Disease | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for ApoE status CSF with Alzheimer markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective MCI cohort: EEG with SPR analysis of the group from the study 2011-2013 is evaluated in relation to the status of current cognitive impairment
  Interventions: Diagnostic Test: EEG with SPR analysis
- Prospective MCI cohort: New individuals diagnosed with MCI. EEG with SPR analysis is performed during the diagnostic work-up and evaluated in relation to changes in cognitive status during the following two years.
  Interventions: Diagnostic Test: EEG with SPR analysis

INTERVENTIONS:
Diagnostic Test: EEG with SPR analysis — qEEG with SPR analysis was performed in group 1 during 2011-2013 and in group 2, the same procedure is performed.

SUMMARY:
Multi center study of six Memory Clinics in four Nordic countries in validating a prognostic diagnostic investigation of qEEG in Mild Cognitive Impairment (MCI). The study is in two parts, the first one is a follow up of a previous study conducted in 2011-2013 and the second half is new recruitment with two years follow up. End points are diagnosis of a dementing disorder, primarily dementia of Alzheimer´s type.

DETAILED DESCRIPTION:
The Nordic Network in Dementia Diagnostics (NIDD) conducted a study in 2011-2013 on qEEG using a method of Statistical Pattern Recognition (SPR) in six academic Memory Clinics in four Nordic countries. In the current study, those from the former study diagnosed either with Mild Cognitive Impairment (MCI; n= 120) or with Subjective Cognitive Impairment (SCI; n=60) are contacted again and evaluated for cognitive impairment. The EEG registered at entry in the former study is considered in relation to their current diagnosis (SCI,MCI or dementia) and thereby, the prognostic value of the method is evaluated.

In the second part of the study (n=120), new patients evaluated in the Memory Clinics and diagnosed with MCI (not SCI) are invited to participate for a two year follow up.

In the diagnostic work-up, simple screening tests and information from a close relative form the basis of the cognitive status (SCI;MCI, Dementia). In evaluating the cause of cognitive impairment, detailed neuropsychological testing is performed as well as MRI of the brain and CSF for Alzheimer´s markers. qEEG with SPR analysis is registered but the clinician is blinded to its outcome.

The end point in both parts of the study is a diagnosis of a dementing disorder.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Individuals diagnosed with either SCI or MCI during 2011-2013 Group 2: Individuals diagnosed with MCI at entry of the study

-

Exclusion Criteria:

* Age <50 years or >85 years
* Medically or psychologically unstable
* Living outside the capital region

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals referred for diagnostic evaluation to an academic Memory Clinic (MC) in either of the six participating centers.
  Group 1: Individuals diagnosed with either SCI or MCI in a study by the same centers in 2011-2013 Group 2: Individuals referred to the same academic MC, diagnosed with the cognitive status of MCI at the first visit. They are followed up for 2 years for evaluation of their cognitive status and if diagnosed with dementia, their disorder is registered.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of dementia | Group 1: 4-6 years after initial registration, Group 2: 1-2 years after initial registration
  The type of dementia is registered

SECONDARY OUTCOMES:
CERAD ten word test | Group 1: 4-6 years after initial registration, Group 2: 1-2 years after initial registration
  Immediate recall (0-30 words); delayed recall (0-10words) and recognition (0-20 words)

CONTACTS AND LOCATIONS:
Overall Officials: Knut Engedal, PhD, Study Director — Ullevaal University Hospital. Oslo, Norway
Locations (1):
- Landspitali University Hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No